CLINICAL TRIAL: NCT01047579
Title: A 12 Week, Multicenter, Open Label Evaluation of Caregiver Preference, Safety and Tolerability of Exelon® Patch (Rivastigmine Transdermal) in Patients With Alzheimer's Disease
Acronym: BETTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CENA713DIL01
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2012-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Rivastigmine transdermal; caregiver preference
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- Rivastigmine transdermal (Other)
  Interventions: Drug: Rivastigmine transdermal

INTERVENTIONS:
Drug: Rivastigmine transdermal

SUMMARY:
This study is designed to evaluate caregiver preference for Exelon® patch (target patch size 10 cm²) treatment in patients with Alzheimer's disease (MMSE 10-26) who were under cholinesterase inhibitor treatment and experienced adverse event/s in a community setting.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease according to the NINCDS-ADRDA and DSM-IV criteria.
* MMSE score of >10 and <26.
* Patients who were under ChE inhibitor treatment and experienced adverse events.
* Residing with someone in the communities throughout the study or if, living alone, in contact with the responsible caregiver every day, primary caregiver willing to accept responsibility for supervising the treatment and condition of the patient.

Exclusion Criteria:

* Involved in other clinical trials or treated by experimental drug within the previous 4 weeks.
* Current diagnosis of an active skin lesion that would prevent accurate assessment of the adhesion and potential skin irritation of the patch.
* History of allergy to topical products containing any of the constitution of the patches.
* Patients with evidence of severe or unstable physical illness, i.e., acute and severe asthmatic conditions, severe or unstable cardiovascular disorders, etc.
* Patients with bradycardia (bpm less than 50) or sick sinus syndrome or conduction defects (sino-atrial block, second degree A-V blocks).
* Patients with body weight less than 40 kg.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Caregiver questionnaire | 12 weeks

SECONDARY OUTCOMES:
Safety and Tolerability. Safety assessments include vital signs and adverse events (AEs) | every visit

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Israel (5):
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigational Site, Haifa
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv